CLINICAL TRIAL: NCT01936519
Title: A Randomized Prospective Trial of Conversion to Everolimus Therapy From Calcineurin Inhibitor Based Maintenance Immunosuppression in Association With Mycophenolic Acid in Liver Transplantation: Examination of Impact on Long Term Renal Function.
Brief Title: Conversion to Everolimus From Calcineurin Inhibitor With Mycophenolic Acid: Impact on Long Term Renal Function in Liver Transplantation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Zakiyah Kadry, Professor of Surgery; Chief, Division of Transplantation, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 38115
Record Dates: First submitted 2013-08-16; First posted 2013-09-06 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Immunosuppression; Renal Failure
Keywords: Everolimus; Zortress; Renal Function; Tacrolimus; Cyclosporine; Myfortic; Mycophenolic Acid; Liver Transplantation
MeSH Terms: conditions — Renal Insufficiency | interventions — Everolimus; Mycophenolic Acid; Calcineurin Inhibitors; Tacrolimus; Cyclosporine; Cyclosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcineurin Inhibitor with Mycophenolic Acid (Active Comparator): Calcineurin inhibitor immunosuppression with mycophenolic acid
  Interventions: Drug: Calcineurin Inhibitor
- Everolimus with Mycophenolic Acid (Experimental): Conversion to Everolimus immunosuppression combined with mycophenolic acid (Myfortic: MPA), and complete discontinuation of Calcineurin inhibitor at 3 months post transplant.
  Interventions: Drug: Arm A: Everolimus

INTERVENTIONS:
Drug: Arm A: Everolimus — Conversion to Everolimus immunosuppression combined with mycophenolic acid (Myfortic: MPA), and complete discontinuation of Calcineurin inhibitor at 3 months post transplant.
  Other Names: Zortress; Mycophenolic Acid (Myfortic)
  Arms: Everolimus with Mycophenolic Acid
Drug: Calcineurin Inhibitor — Comparison Arm: Continuation with standard immunosuppressive therapy consisting of Calcineurin inhibitor associated with mycophenolic acid (Myfortic: MPA).
  Other Names: Tacrolimus (Prograf); Cyclosporine (Gengraf); Mycophenolic Acid (Myfortic)
  Arms: Calcineurin Inhibitor with Mycophenolic Acid

SUMMARY:
This study will examine the renal sparing impact of implementing a strategy of conversion to everolimus from a calcineurin inhibitor based immunosuppressive protocol at 3 months post liver transplant

DETAILED DESCRIPTION:
Given the increasing proportion of patients having renal failure at the time of transplant, with the nephrotoxic effect of calcineurin inhibitor based immunosuppression associated with its long term negative survival impact, this study proposes to examine the renal sparing impact of conversion to everolimus from a calcineurin inhibitor based immunosuppressive protocol at 3 months post liver transplant. The 3 month time point was chosen to allow for the switch to everolimus to occur at a period of stable post transplant liver function when both technical and rejection risks are lower. The 3 month cut off was also chosen because of data indicating that worsening renal function at 4 weeks, 3 months and 1 year post transplant is an independent risk factor for the development of chronic renal failure and end stage renal disease after orthotopic liver transplantation. 24 patients will be randomized into 2 arms:

Arm A: Conversion to Everolimus immunosuppression combined with mycophenolic acid (Myfortic: MPA), and complete discontinuation of Calcineurin inhibitor at 3 months post transplant.

Arm B: Continuation with standard immunosuppressive therapy consisting of Calcineurin inhibitor associated with mycophenolic acid (Myfortic: MPA).

Follow up: 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to provide written informed consent and adhere to study regimen.
* Primary deceased donor liver transplant recipients 18-70 years of age
* Functioning allograft at randomization (AST, ALT, Total Bilirubin levels ≤3 times ULN, and AlkP and GGT levels ≤ 5 times ULN). Elevated GGT alone, in combination with AST, ALT, total bilirubin and AlkP within defined range does not exclude patients from randomization.
* Recipients on an immunosuppressive regimen of corticosteroids and tacrolimus.
* Confirmed recipient HCV status at Screening (either by serology or PCR).
* Abbreviated MDRD eGFR ≥ 30 mL/min/1.73m2. Local and central serum creatinine results within 5 days prior to randomization, however no sooner than Day 25 post-transplantation.
* Verification of at least one tacrolimus trough level of ≥ 8 ng/mL one week prior to randomization. Target trough levels above 8 ng/mL prior to randomization.
* Patients able to take oral medication at time of randomization.

Exclusion Criteria:

* Recipients of multiple solid organ or islet cell tissue transplants, or have previously received an organ or tissue transplant. Combined liver kidney transplant recipients.
* Living donor or split liver recipients.
* History of malignancy of any organ system within past 5 years whether or not there is evidence of local recurrence or metastases, other than non-metastatic basal or squamous cell carcinoma of the skin or HCC.
* Hepatocellular carcinoma that does not fulfill Milan criteria (1 nodule ≤ 5 cm, 2-3 nodules all < 3 cm, per explant histology of recipient liver.
* Use of antibody induction therapy.
* Patients with known hypersensitivity to the drugs used on study or their class, or to any of the excipients.
* Recipients of ABO incompatible transplant grafts.
* Recipients of Hepatitis B surface antigen or HIV donor organs.
* Surgical or medical condition, which might significantly alter absorption, distribution, metabolism and excretion of study drug.
* Women of child-bearing potential (WOCBP): all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS (1) they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/m, or (2) have past 6 weeks from surgical bilateral oophorectomy with or without hysterectomy or (3) are using one or more of the following methods of contraception: surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), copper coated IUD and double-barrier methods ( any double combination of male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception should be maintained throughout and for 3 months after study drug discontinuation.
* History of coagulopathy or medical condition requiring long-term anticoagulation which would preclude liver biopsy after transplantation. (Low dose aspirin treatment or interruption of chronic anticoagulant is allowed).

Enrollment Exclusion - Randomization

* Severe hypercholesterolemia (>350 mg/dL; >9 mmol/L) or hypertriglyceridemia (>500 mg/dL; >8.5 mmol/L) within 6 months of transplantation. Controlled hyperlipidemia is acceptable at time of randomization.
* Platelet count < 50,000/mm3 at randomization.
* Absolute neutrophil count < 1,000/mm³ or white blood cell count <2,000/mm³ at randomization.
* Patients positive for HIV: Negative laboratory results within 6 months before randomization are acceptable.
* Clinically significant systemic infection requiring IV antibiotics at randomization. Patients in a critical care setting at randomization requiring life support measures such as mechanical ventilation, dialysis, or vasopressor agents.
* Patients on renal replacement therapy within 7 days prior to randomization.
* Thrombosis of major hepatic arteries, major hepatic veins, portal vein and inferior vena cava. Results obtained within 5 days prior to randomization are acceptable, however no sooner than Day 25 post-transplantation.
* Acute rejection requiring antibody therapy or more than one steroid sensitive episode of acute rejection during the run-in period. Includes patients who have not completed steroid treatment for acute rejection within 7 days prior to randomization.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zakiyah Kadry, MD, Principal Investigator — Penn State College of Medicine; Penn State Milton S Hershey Medical Center
Locations (1):
- Penn State College of Medicine; Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to publish de-identified data

REFERENCES:
- [Background] Burra P, Senzolo M, Masier A, Prestele H, Jones R, Samuel D, Villamil F. Factors influencing renal function after liver transplantation. Results from the MOST, an international observational study. Dig Liver Dis. 2009 May;41(5):350-6. doi: 10.1016/j.dld.2008.09.018. Epub 2008 Nov 28. PMID 19046932
- [Background] Gonwa TA, Mai ML, Melton LB, Hays SR, Goldstein RM, Levy MF, Klintmalm GB. End-stage renal disease (ESRD) after orthotopic liver transplantation (OLTX) using calcineurin-based immunotherapy: risk of development and treatment. Transplantation. 2001 Dec 27;72(12):1934-9. doi: 10.1097/00007890-200112270-00012. PMID 11773892
- [Background] Ojo AO, Held PJ, Port FK, Wolfe RA, Leichtman AB, Young EW, Arndorfer J, Christensen L, Merion RM. Chronic renal failure after transplantation of a nonrenal organ. N Engl J Med. 2003 Sep 4;349(10):931-40. doi: 10.1056/NEJMoa021744. PMID 12954741
- [Background] Velidedeoglu E, Bloom RD, Crawford MD, Desai NM, Campos L, Abt PL, Markmann JW, Mange KC, Olthoff KM, Shaked A, Markmann JF. Early kidney dysfunction post liver transplantation predicts late chronic kidney disease. Transplantation. 2004 Feb 27;77(4):553-6. doi: 10.1097/01.tp.0000114609.99558.41. PMID 15084934
- [Background] Wadei HM, Geiger XJ, Cortese C, Mai ML, Kramer DJ, Rosser BG, Keaveny AP, Willingham DL, Ahsan N, Gonwa TA. Kidney allocation to liver transplant candidates with renal failure of undetermined etiology: role of percutaneous renal biopsy. Am J Transplant. 2008 Dec;8(12):2618-26. doi: 10.1111/j.1600-6143.2008.02426.x. PMID 19032225
- [Background] Randhawa PS, Shapiro R. Chronic renal failure after liver transplantation. Am J Transplant. 2005 May;5(5):967-8. doi: 10.1111/j.1600-6143.2005.00819.x. No abstract available. PMID 15816874
- [Background] McCauley J, Van Thiel DH, Starzl TE, Puschett JB. Acute and chronic renal failure in liver transplantation. Nephron. 1990;55(2):121-8. doi: 10.1159/000185938. PMID 2362625
- [Background] Fisher NC, Nightingale PG, Gunson BK, Lipkin GW, Neuberger JM. Chronic renal failure following liver transplantation: a retrospective analysis. Transplantation. 1998 Jul 15;66(1):59-66. doi: 10.1097/00007890-199807150-00010. PMID 9679823
- [Background] Neuberger JM, Mamelok RD, Neuhaus P, Pirenne J, Samuel D, Isoniemi H, Rostaing L, Rimola A, Marshall S, Mayer AD; ReSpECT Study Group. Delayed introduction of reduced-dose tacrolimus, and renal function in liver transplantation: the 'ReSpECT' study. Am J Transplant. 2009 Feb;9(2):327-36. doi: 10.1111/j.1600-6143.2008.02493.x. Epub 2008 Dec 15. PMID 19120077
- [Background] Chapman TM, Perry CM. Everolimus. Drugs. 2004;64(8):861-72; discussion 873-4. doi: 10.2165/00003495-200464080-00005. PMID 15059040
- [Background] Levy G, Schmidli H, Punch J, Tuttle-Newhall E, Mayer D, Neuhaus P, Samuel D, Nashan B, Klempnauer J, Langnas A, Calmus Y, Rogiers X, Abecassis M, Freeman R, Sloof M, Roberts J, Fischer L. Safety, tolerability, and efficacy of everolimus in de novo liver transplant recipients: 12- and 36-month results. Liver Transpl. 2006 Nov;12(11):1640-8. doi: 10.1002/lt.20707. PMID 16598777
- [Background] Nashan B. Early clinical experience with a novel rapamycin derivative. Ther Drug Monit. 2002 Feb;24(1):53-8. doi: 10.1097/00007691-200202000-00010. PMID 11805723
- [Background] Chan L, Greenstein S, Hardy MA, Hartmann E, Bunnapradist S, Cibrik D, Shaw LM, Munir L, Ulbricht B, Cooper M; CRADUS09 Study Group. Multicenter, randomized study of the use of everolimus with tacrolimus after renal transplantation demonstrates its effectiveness. Transplantation. 2008 Mar 27;85(6):821-6. doi: 10.1097/TP.0b013e318166927b. PMID 18360262
- [Background] Everson GT. Everolimus and mTOR inhibitors in liver transplantation: opening the "box". Liver Transpl. 2006 Nov;12(11):1571-3. doi: 10.1002/lt.20845. No abstract available. PMID 17058246
- [Background] De Simone P, Carrai P, Precisi A, Petruccelli S, Baldoni L, Balzano E, Ducci J, Caneschi F, Coletti L, Campani D, Filipponi F. Conversion to everolimus monotherapy in maintenance liver transplantation: feasibility, safety, and impact on renal function. Transpl Int. 2009 Mar;22(3):279-86. doi: 10.1111/j.1432-2277.2008.00768.x. Epub 2008 Dec 2. PMID 19054383
- [Background] Johnson RW, Kreis H, Oberbauer R, Brattstrom C, Claesson K, Eris J. Sirolimus allows early cyclosporine withdrawal in renal transplantation resulting in improved renal function and lower blood pressure. Transplantation. 2001 Sep 15;72(5):777-86. doi: 10.1097/00007890-200109150-00007. PMID 11571437
- [Background] Oberbauer R, Segoloni G, Campistol JM, Kreis H, Mota A, Lawen J, Russ G, Grinyo JM, Stallone G, Hartmann A, Pinto JR, Chapman J, Burke JT, Brault Y, Neylan JF; Rapamune Maintenance Regimen Study Group. Early cyclosporine withdrawal from a sirolimus-based regimen results in better renal allograft survival and renal function at 48 months after transplantation. Transpl Int. 2005 Jan;18(1):22-8. doi: 10.1111/j.1432-2277.2004.00052.x. PMID 15612979
- [Background] Ekberg H. Calcineurin inhibitor sparing in renal transplantation. Transplantation. 2008 Sep 27;86(6):761-7. doi: 10.1097/TP.0b013e3181856f39. PMID 18813097
- [Background] Baboolal K. A phase III prospective, randomized study to evaluate concentration-controlled sirolimus (rapamune) with cyclosporine dose minimization or elimination at six months in de novo renal allograft recipients. Transplantation. 2003 Apr 27;75(8):1404-8. doi: 10.1097/01.TP.0000063703.32564.3B. PMID 12717239
- [Background] Webster AC, Lee VW, Chapman JR, Craig JC. Target of rapamycin inhibitors (sirolimus and everolimus) for primary immunosuppression of kidney transplant recipients: a systematic review and meta-analysis of randomized trials. Transplantation. 2006 May 15;81(9):1234-48. doi: 10.1097/01.tp.0000219703.39149.85. PMID 16699448
- [Background] Eisen HJ, Tuzcu EM, Dorent R, Kobashigawa J, Mancini D, Valantine-von Kaeppler HA, Starling RC, Sorensen K, Hummel M, Lind JM, Abeywickrama KH, Bernhardt P; RAD B253 Study Group. Everolimus for the prevention of allograft rejection and vasculopathy in cardiac-transplant recipients. N Engl J Med. 2003 Aug 28;349(9):847-58. doi: 10.1056/NEJMoa022171. PMID 12944570
- [Background] Levy GA, Grant D, Paradis K, Campestrini J, Smith T, Kovarik JM. Pharmacokinetics and tolerability of 40-0-[2-hydroxyethyl]rapamycin in de novo liver transplant recipients. Transplantation. 2001 Jan 15;71(1):160-3. doi: 10.1097/00007890-200101150-00028. PMID 11211186
- [Background] Gomez-Camarero J, Salcedo M, Rincon D, Lo Iacono O, Ripoll C, Hernando A, Sanz C, Clemente G, Banares R. Use of everolimus as a rescue immunosuppressive therapy in liver transplant patients with neoplasms. Transplantation. 2007 Sep 27;84(6):786-91. doi: 10.1097/01.tp.0000280549.93403.dd. PMID 17893613
- [Background] Yu SF, Wu LH, Zheng SS. Genetic factors for individual administration of immunosuppressants in organ transplantation. Hepatobiliary Pancreat Dis Int. 2006 Aug;5(3):337-44. PMID 16911928
- [Background] Chaudhary MA, Stearns SC. Estimating confidence intervals for cost-effectiveness ratios: an example from a randomized trial. Stat Med. 1996 Jul 15;15(13):1447-58. doi: 10.1002/(SICI)1097-0258(19960715)15:133.0.CO;2-V. PMID 8841654
- [Background] Willan AR, O'Brien BJ. Confidence intervals for cost-effectiveness ratios: an application of Fieller's theorem. Health Econ. 1996 Jul-Aug;5(4):297-305. doi: 10.1002/(SICI)1099-1050(199607)5:43.0.CO;2-T. PMID 8880166
- [Background] Briggs AH, Wonderling DE, Mooney CZ. Pulling cost-effectiveness analysis up by its bootstraps: a non-parametric approach to confidence interval estimation. Health Econ. 1997 Jul-Aug;6(4):327-40. doi: 10.1002/(sici)1099-1050(199707)6:43.0.co;2-w. PMID 9285227
- [Background] Lothgren M, Zethraeus N. Definition, interpretation and calculation of cost-effectiveness acceptability curves. Health Econ. 2000 Oct;9(7):623-30. doi: 10.1002/1099-1050(200010)9:73.0.co;2-v. PMID 11103928
- [Background] Fairbanks KD, Eustace JA, Fine D, Thuluvath PJ. Renal function improves in liver transplant recipients when switched from a calcineurin inhibitor to sirolimus. Liver Transpl. 2003 Oct;9(10):1079-85. doi: 10.1053/jlts.2003.50183. PMID 14526403

RESULTS

PARTICIPANT FLOW:
Groups:
- Calcineurin Inhibitor and Mycophenolic Acid: Calcineurin inhibitor immunosuppression with mycophenolic acid
  Calcineurin Inhibitor: Comparison Arm: Continuation with standard immunosuppressive therapy consisting of Calcineurin inhibitor associated with mycophenolic acid (Myfortic: MPA).
- Everolimus and Mycophenolic Acid: Conversion to Everolimus immunosuppression combined with mycophenolic acid (Myfortic: MPA), and complete discontinuation of Calcineurin inhibitor at 3 months post transplant.
  Everolimus: Conversion to Everolimus immunosuppression combined with mycophenolic acid (Myfortic: MPA), and complete discontinuation of Calcineurin inhibitor at 3 months post transplant.
Period: Overall Study
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid
Started | 12 | 12
Completed | 11 | 8
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Full Range); unit: years] | 55.1 [45 to 69] | 56.5 [37 to 70] | 55.79 [37 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 10 | 11 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
Serum Creatinine [Mean (Full Range); unit: mg/dL] | 1.3 [0.79 to 1.78] | 1.23 [0.62 to 1.8] | 1.26 [0.62 to 1.8]
Cockcroft Gault Creatinine Clearance [Mean (Full Range); unit: ml/min] | 78.11 [42.48 to 144.58] | 85.15 [44.27 to 175.99] | 81.63 [42.48 to 175.99]
Modification of Diet in Renal Disease (MDRD) Clearance [Mean (Full Range); unit: mL/min/1.73 m^2] | 61.24 [40 to 108.12] | 69.91 [38.2 to 140.92] | 65.58 [38.2 to 140.92]
24 Hour Urine Creatinine Clearance [Mean (Full Range); unit: mL/min/1.73m2] | 64 [17 to 200] | 59.25 [24 to 99] | 61.63 [17 to 200]
Iothalamate Clearance [Mean (Full Range); unit: ml/min] | 60.60 [16.14 to 141.54] | 58.10 [31.46 to 110.63] | 59.35 [16.14 to 141.54]
24hr Urine Protein [Mean (Full Range); unit: g/24hrs] | 0.2 [0.039 to 0.504] | 0.19 [0.055 to 0.52] | 0.1925 [0.039 to 0.52]

OUTCOME MEASURES:

1. Primary Outcome: Renal Function as Measured by 24 Hour Urine Creatinine Clearance
Description: Renal Function was assessed by 24 hr urine collection creatinine clearance measured (mL/min). 24 Hr urine collection was assessed at baseline, 6 months, 1 year, and 2 years post transplant.
Time Frame: 6 months, 1 year, and 2 years
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Calcineurin Inhibitor With Mycophenolic Acid | Everolimus With Mycophenolic Acid
Number analyzed (Participants) | 11 | 8
mL/min
  24hr Urine Creatinine Clearance at 6 months | 68.09 (30.08) | 70.75 (29.03)
  24hr Urine Creatinine Clearance at 1 year | 68.09 (28.91) | 86.8 (29.34)
  24hr Urine Creatinine Clearance at 2 years | 61.54 (27.5) | 90.63 (30.05)

2. Primary Outcome: Renal Function as Measured by Serum Creatinine Level
Description: Serum creatinine levels were assessed at 6 months, 1 year, and 2 years post transplant
Time Frame: 6 months, 1 year, and 2 years
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid
Number analyzed (Participants) | 11 | 8
mg/dL
  Serum Creatinine at 6 months | 1.29 (0.43) | 1.02 (0.24)
  Serum Creatinine at 1 year | 1.29 (0.38) | 0.95 (0.25)
  Serum Creatinine at 2 years | 1.51 (0.69) | 0.95 (0.30)

3. Primary Outcome: Renal Function as Measured by Cockcroft Gault Creatinine Clearance
Description: The Cockcroft-Gault formula for estimating creatinine clearance was determined at 6 months, 1 year, and 2 years post transplant
Time Frame: 6 months, 1 year, and 2 years
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid
Number analyzed (Participants) | 11 | 8
mL/min/1.73m2
  Cockcroft Gault Creatinine Clearance at 6 months | 79.84 (29.29) | 100.17 (45.39)
  Cockcroft Gault Creatinine Clearance at 1 year | 86.84 (37.17) | 113.47 (60.76)
  Cockcroft Gault Creatinine Clearance at 2 years | 80.85 (28.57) | 108.16 (60.1)
Statistical Analysis 1: Comparison: Calcineurin Inhibitor and Mycophenolic Acid vs Everolimus and Mycophenolic Acid; Statistical analysis was performed on the Cockcroft Gault Creatinine clearance 2 year data; Test type: Equivalence — Mann Whitney U Test was performed; p = 0.283, Wilcoxon (Mann-Whitney) — Cockcroft-Gault Clearance; Mean Difference (Net) = 27.32, 95% CI 2-sided [-16.17 to 70.80], Standard Error of Mean 20.61

4. Primary Outcome: Renal Function as Measured by Modification of Diet in Renal Disease (MDRD) Estimated Glomerular Filtration Rate (eGFR)
Description: Modification of Diet in Renal Disease (MDRD) estimated Glomerular Filtration Rate (eGFR) was assessed at 6 months, 1 year, and 2 years post transplant.
Time Frame: 6 months, 1 year, and 2 years
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m2
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid
Number analyzed (Participants) | 11 | 8
mL/min/1.73 m2
  MDRD eGFR at 6 months | 62.18 (22.51) | 81.27 (31.30)
  MDRD eGFR at 1 year | 60.63 (19.68) | 88.01 (34.08)
  MDRD eGFR at 2 years | 53.29 (17.58) | 87.37 (32.09)
Statistical Analysis 1: Comparison: Calcineurin Inhibitor and Mycophenolic Acid vs Everolimus and Mycophenolic Acid; Statistical analysis was performed on the MDRD Clearance 2 year data row data; Test type: Equivalence — Wilcoxon Test; p = 0.013, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 34.08, 95% CI 2-sided [9.95 to 58.21], Standard Error of Mean 11.44

5. Primary Outcome: Renal Function as Measured by Iothalamate Clearance
Description: Iothalamate Clearance was assessed at 6 months, 1 year, and 2 years post transplant.
Time Frame: 6 months, 1 year, and 2 years
Measure: Mean (Standard Deviation); unit: mL/min/1.73m2
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid
Number analyzed (Participants) | 11 | 8
mL/min/1.73m2
  Iothalamate Clearance at 6 months | 67.99 (39.23) | 74.23 (31.30)
  Iothalamate Clearance at 1 year | 66.65 (32.69) | 104.01 (43)
  Iothalamate Clearance at 2 years | 57.19 (24.75) | 79.41 (27.71)
Statistical Analysis 1: Comparison: Calcineurin Inhibitor and Mycophenolic Acid vs Everolimus and Mycophenolic Acid; Statistical analysis was performed on the Iothalamate Clearance 2 year data; Test type: Equivalence — Wilcoxon Test; p = 0.099, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 22.22, 95% CI 2-sided [-3.28 to 47.72], Standard Error of Mean 12.09
Statistical Analysis 2: Comparison: Everolimus and Mycophenolic Acid; Power and sample size. The assumption was made that eGFR would improve from 34 mL/min/1.73 m2 to 43 mL/min/1.73 m2. It was determined that a sample size of 12 in each group would have 80% power to detect a difference in means of -9.0 (the difference between a group 1 mean of 34.0 and a group 2 mean of 43.0) assuming that the common standard deviation was 7.5 using a two group t-test with a 0.05 two-sided significance level. Data from the 2 year time point was used for analysis; Test type: Equivalence — Non-parametric statistical tests were used for all analyses, including the Mann-Whitney U test for continuous outcomes and Pearson's chi-square test for binary outcomes. Univariate statistical tests were used for all comparisons. Cohen's d was utilized for all comparisons to provide information about effect size; p = .032, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 29.08, 95% CI 2-sided [1.04 to 57.1], Standard Error of Mean 13.29
Statistical Analysis 3: Comparison: Calcineurin Inhibitor and Mycophenolic Acid vs Everolimus and Mycophenolic Acid; Statistical analysis was performed on 2 year data time point; Test type: Equivalence — Difference of zero hypothesized; p = 0.015, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-1.11 to -0.003], Standard Error of Mean 0.263

6. Other Pre Specified Outcome: Recipient and Donor Genotyping for Selected Variants of CYP3A5, ABCB1 (MDR1), and CYP4A Genes
Description: A blood sample was obtained from recipients and donors to measure gene polymorphism effects on metabolism of calcineurin inhibitor and everolimus. The polymorphisms are represented as the number of SNP occurrences for the CYP3A5, ABCB1 (MDR1) gene, and CYP4A4*22 genes.
Time Frame: 2 years
Population: SNP source: rs776746 = CYP3A5 gene; rs1045642, rs1128503 and rs2032582 = ABCB1 (MDR1) gene, and rs35599367=Cyp4A4*22 gene.
Measure: Count of Participants; unit: Participants
Groups:
- Everolimus and Mycophenolic Acid: Conversion to Everolimus immunosuppression combined with mycophenolic acid (Myfortic: MPA), and complete discontinuation of Calcineurin inhibitor at 3 months post transplant.
  Arm A: Everolimus: Conversion to Everolimus immunosuppression combined with mycophenolic acid (Myfortic: MPA), and complete discontinuation of Calcineurin inhibitor at 3 months post transplant.
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid
Number analyzed (Participants) | 11 | 11
Participants
  Recipient Genotypes : rs776746 (CYP3A5 gene) | 11 | 11
  Recipient Genotypes : rs1045642 (ABCB1 gene) | 6 | 6
  Recipient Genotypes : rs1128503 (ABCB1 gene) | 7 | 8
  Recipient Genotypes : rs2032582 (ABCB1 gene) | 1 | 0
  Recipient Genotypes : rs35599367 (CYP4A4*22 gene) | 1 | 1
  Donor Genotypes : rs776746 (CYP3A5 gene) | 3 | 0
  Donor Genotypes : rs1045642 (ABCB1 gene) | 1 | 5
  Donor Genotypes : rs1128503 (ABCB1 gene) | 0 | 0
  Donor Genotypes : rs2032582 (ABCB1 gene) | 0 | 0
  Donor Genotypes : rs35599367 (Cyp4A4*22) | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Calcineurin Inhibitor and Mycophenolic Acid | Everolimus and Mycophenolic Acid
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcineurin Inhibitor and Mycophenolic Acid (N=12) | Everolimus and Mycophenolic Acid (N=12)
Hepatic Artery Thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Subject was found to have incidentally a hepatic artery thrombosis at 6 months on a CT scan for tumor screening. Liver function tests were normal and patient was asymptomatic.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcineurin Inhibitor and Mycophenolic Acid (N=12) | Everolimus and Mycophenolic Acid (N=12)
Leukopenia (Immune system disorders) | 7 (7) | 9 (9) — Low white cell count
Hyperlipidemia (Metabolism and nutrition disorders) | 7 (7) | 9 (9) — Hyperlipidemia requiring treatment
Cellular Rejection (Immune system disorders) | 1 (1) | 3 (3) — T-cell mediated liver organ rejection
antibody mediated rejection (Immune system disorders) | 1 (1) | 2 (2) — Donor specific antibody positive level.
Cytomegalovirus Infection (Infections and infestations) | 6 (6) | 2 (2)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1) — Hepatitis c infection recurrence after liver transplantation
Minor Infection (Infections and infestations) | 3 (3) | 5 (5) — Minor infections includes: ascites infection, upper respiratory infection, sinusitis, fever, cholangitis, cold/flu.
Dental Infection (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Difficile (Infections and infestations) | 1 (1) | 0 (0)
Herpes Simplex & Zoster (Infections and infestations) | 1 (1) | 2 (2)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Hypertension (General disorders) | 4 (4) | 3 (3)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Pulmonary hypertension of unknown cause. Treated.
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 1 (1) — Depression requiring treatment &/or psychiatric evaluation
Temor (Nervous system disorders) | 1 (1) | 0 (0) — Tremor of the upper extremities
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5) | 1 (1) — Low serum magnesium requiring correction
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Low serum calcium level
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Low serum potassium level
hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — High serum glucose level
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) — High serum potassium level requiring correction/treatment
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 2 (2) — Edema of the lower extremities and increased weight due to fluid retention
skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) — Squamous and/or basal cell skin cancer
Hepatic Steatosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Fatty liver
Low Serum Testosterone Level (Reproductive system and breast disorders) | 3 (3) | 5 (5) — Serum Testosterone level was measured at baseline, 6, 12 & 24 months. Was significantly lower at 6 & 12 months in the Everolimus arm and showed a lower trend at 24 months.
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Emesis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper Gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — Upper gastrointestinal bleeding from duodenal arterio-venous malformation
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT01936519/Prot_SAP_000.pdf